CLINICAL TRIAL: NCT04180982
Title: A Phase II, MultiCenter, Double-Blind Study to Evaluate the Efficacy and Safety of SHR4640 and Febuxostat in Subjects With Hyperuricemia
Brief Title: A Safety and Efficacy Study of SHR4640 and Febuxostat in Subjects With Hyperuricemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR4640-202
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental): SHR4640 dose1 Oral Tablet plus Febuxostat dose1 Oral Tablet Day1~Day28 qd.
  Interventions: Drug: SHR4640 dose1 plus Febuxostat dose1
- Treatment group B (Experimental): SHR4640 dose1 Oral Tablet plus Febuxostat dose2 Oral Tablet Day1~Day28 qd.
  Interventions: Drug: SHR4640 dose1 plus Febuxostat dose2
- Treatment group C (Experimental): SHR4640 dose2 Oral Tablet plus Febuxostat dose3 Oral Tablet Day1~Day28 qd.
  Interventions: Drug: SHR4640 dose2 plus Febuxostat dose3

INTERVENTIONS:
Drug: SHR4640 dose1 plus Febuxostat dose1 — Tablet,dose1,QD
  Arms: Treatment group A
Drug: SHR4640 dose1 plus Febuxostat dose2 — Tablet,dose1, dose2 QD
  Arms: Treatment group B
Drug: SHR4640 dose2 plus Febuxostat dose3 — Tablet,dose2, dose3 QD
  Arms: Treatment group C

SUMMARY:
The objective of the study is to assess the Safety and Efficacy of SHR4640 and Febuxostat in patients with Hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index ≥18 and ≤30 kg/m2;
* Screening sUA value ≥8mg/dl;
* Subject has no clinically relevant abnormalities in vital signs, ECG, physical examination，imaging examination or safety laboratory values.

Exclusion Criteria:

* Subject known or suspected of being sensitive to the study drugs or its ingredient；
* ALT、AST、TBIL>1.5ULN;
* History of kidney stones or screening kidney stones by B-ultrasound；
* History of malignancy；
* History of xanthinuria；
* Donated blood（≥400ml）within 3 months prior to screening or received transfusion of blood.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-12-03 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events(AEs) and Serious Adverse Events(SAEs) | Up to week 4
  Incidence of AEs and SAEs, incidence of Treatment-Emergent Adverse Events, incidence of drug related adverse events (safety and tolerability)

SECONDARY OUTCOMES:
Percentage of subjects with a serum uric level≤360μmol/L | At week1, 2, 3 and 4
Percentage change from baseline in serum uric level . | At week1, 2, 3 and 4
Actual change from baseline in serum uric level | At week1, 2, 3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Liu Yi, Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: No